CLINICAL TRIAL: NCT00568165
Title: Value of a Mobile Team of Cardiologist Using Echocardiography for Managing Patients With Acute Heart Failure
Brief Title: EMEPIC : Value of a Mobile Team of Cardiologist Using Echocardiography for Managing Patients With Acute Heart Failure
Acronym: EMEPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Paris 7 - Denis Diderot (Other)
Responsible Party: Pr. Guillaume JONDEAU, University Paris 7
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Code IDRCD : 2007- A00640 - 53; N°CPP : 0711602; N°CCTIRS : 07331
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Last update posted 2010-10-26 (Estimated); Status verified 2010-08

CONDITIONS: Acute Heart Failure; Congestive Edema; Cardiac Disease
Keywords: Heart failure, congestive; Echocardiography; Patient care team
MeSH Terms: conditions — Heart Diseases; Heart Failure | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Mobile Team
  Interventions: Procedure: Mobile team
- 2 (Active Comparator): Standard care
  Interventions: Procedure: Standard care

INTERVENTIONS:
Procedure: Mobile team — a mobile team including a cardiologist with mobile echocardiography, systematic follow up à 3 days, a dietician advice in patients hospitalized for acute heart failure in a non cardiology ward
  Arms: 1
Procedure: Standard care — Standard care
  Arms: 2

SUMMARY:
The aim of the study is to compare clinical management of patients with acute decompensation of heart failure, hospitalized in non cardiological ward, with the use of a mobile team including a cardiologist with portable echocardiography and standard care. The hypothesis is that a mobile team will lead to shorter hospitalization.

DETAILED DESCRIPTION:
Randomized, controlled, monocentric study comparing Standard care with the care provided by a mobile team including a cardiologist with mobile echocardiography, systematic follow up à 3 days, a dietician advice in patients hospitalized for acute heart failure in a non cardiology ward on the duration of hospitalization, re-hospitalization rate à 30 days, emergency visit within 30 days, treatment at discharge, mortality within hospital stay and at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized for suspected heart failure
* > or = 18 years

Exclusion Criteria:

* Refuses to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2008-02; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Duration of hospitalization. | 30 days

SECONDARY OUTCOMES:
Re-hospitalization rate à 30 days Emergency visit within 30 days Treatment at discharge Mortality within hospital stay Mortality at 30 days | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume JONDEAU, MD, PhD, Principal Investigator — UNIVERSITY PARIS 7
Locations (1):
- JONDEAU, Paris, France